CLINICAL TRIAL: NCT04845139
Title: A Case Study of Nivolumab for Relapsed/Refractory Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0139
Record Dates: First submitted 2021-04-11; First posted 2021-04-14 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Refractory Central Nervous System Lymphoma; Relapsed Primary Central Nervous System Lymphoma; Primary Central Nervous System Lymphoma
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab administration (Experimental): Nivolumab administration Q2W by intraventricular injection through Ommaya reservoir
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab given intraventricularly
  Other Names: NIVO；Opdivo; BMS-936558

SUMMARY:
The purpose of this study is to determine whether Nivolumab given intrathecally is effective in the treatment of Relapsed/Refractory Primary Central Nervous System Lymphoma (PCNSL)

DETAILED DESCRIPTION:
This is a case study aiming to recruit 1 patient. This study is indicated for relapsed/refractory primary central nervous system lymphoma. Primary objective is to explore the safety.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ECOG 0,1,2,3
* Subjects with pathologically confirmed PCNSL with lesion in brain who progressed after or did not respond to at least 1 line of systemic therapy. PCNSL prior therapy may include HD-MTX, HD-MTX-based regimen, high-dose cytarabine, radiation therapy alone as treatment or as part of consolidation therapy, high-dose therapy with autologous stem cell transplant as part of consolidation therapy, and/or intraocular MTX alone or as part of consolidation therapy
* Subject with sufficient function of liver, kidney, heart, lung and hematopoiesis
* Subjects with relapsed PCNSL and are able to receive biopsy

Exclusion Criteria:

* Subjects that are not DLBCL type pathologically
* Intraocular PCNSL without evidence of brain disease
* Subjects who cannot undergo MRI assessments
* Relapsed PCNSL patients who cannot undergo biopsy
* Biopsy suggests no significant tumor-infiltration T cell or poor PD-1 expression
* Subjects with other malignancy
* Subjects with history of any inflammatory CNS diseases
* Subjects with an active, known, or suspected autoimmune disease
* Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of start of study treatment
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | On a continuous basis up to 1 month after the first dose of study drug
  Adverse events Adverse events assessed according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Best overall response(BOR) | up to 3 months after the first dose of study drug
  Record individual best overall response(BOR), including CR, PR, SD, PD

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Zhang, M.D., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Jianmin Zhang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No